CLINICAL TRIAL: NCT05005520
Title: A Randomized, Double-Blind, Single-Center, Placebo-Controlled Phase 1 Study to Evaluate the Safety, Tolerability, PK and PD of Intravenous DTRI-031 in Healthy Volunteers
Brief Title: Study of DTRI-031 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Basking Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BB-CLIN-101
Record Dates: First submitted 2021-08-09; First posted 2021-08-13 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Healthy Volunteers; Pharmacokinetics; Pharmacodynamics

STUDY DESIGN:
Intervention Model Description: Randomized, placebo-controlled, double-blinded, dose escalation to evaluate the safety, PK, and PD of a single dose of investigational drug or placebo
Who Masked: Participant, Investigator
Masking Description: Double blinded, placebo-controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active Comparator: Single ascending dose DTRI-031 (Active Comparator): Drug: DTRI-031 Single doses of DTRI-031 delivered via intravenous injection. Ascending dose levels will be evaluated.
  Interventions: Drug: DTRI-031
- Placebo Comparator: Single Dose Placebo (Placebo Comparator): Drug: Placebo Single doses of placebo delivered via intravenous injection, matched to DTRI-031 cohorts
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DTRI-031 — Investigational drug
  Arms: Active Comparator: Single ascending dose DTRI-031
Drug: Placebo — Matching placebo to DTRI-031
  Arms: Placebo Comparator: Single Dose Placebo

SUMMARY:
A randomized, double-blind, single center, placebo-controlled phase 1 study in healthy volunteers to assess safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of a single intravenous (iv) injection of DTRI-031

DETAILED DESCRIPTION:
Up to 5 cohorts of 8 healthy volunteers for a total of 40 volunteers will be randomized to either DTRI-031 or matching placebo (6 active:2 placebo). Two sentinel subjects, one randomized to each group, will be dosed at least 1 day prior to dosing of the remaining subjects in a cohort.

Subjects will complete a screening visit up to 28 days prior to administration of study drug to confirm eligibility. Eligible subjects will arrive at the phase 1 unit up to 24 hours prior to Day 1 and remain until completion of 24-hour assessments. Subjects will return for a Day 7 follow-up visit and receive a safety assessment telephone call on Day 28.

A Safety Review Committee will review individual subject and aggregate group safety data following each dose-based study cohort and recommend whether the trial should continue to the next cohort.

ELIGIBILITY:
Inclusion Criteria:

* 18-55 years of age
* Ability to provide written consent
* Weight 50-110 kg with BMI 18.5-32 kg/m2
* Willingness to use contraceptives
* Negative COVID-19 test
* Negative results for alcohol and drugs of abuse

Exclusion Criteria:

* Pregnant or lactating females
* Familial bleeding disorder or individual or family history of bleeding diathesis or coagulopathy
* Females with active menstruation on day of dosing
* Use of prescription medications known to affect platelet function
* Use of NSAIDs, aspirin, anti-platelet or anti-coagulation therapy within 10 days of dosing
* Contraindication to anticoagulation or increased bleeding risks
* History of thrombocytosis, high platelet count, intracranial bleeding, aneurysm, stroke, vascular disease
* History of peptic ulcer disease, gastrointestinal or genitourinary bleed, severe trauma, fracture, major surgery of biopsy of parenchymal organ within past 3 months
* Planned surgery during the study
* Any clinical significant abnormality at screening
* Use of investigational drug in past 30 days or 5 half lives
* Concurrent enrollment in another clinical study or more than 3 clinical studies in past 12 months
* Any prior history of substance abuse or treatment or positive urine screen for drugs of abuse or positive breathalyzer test

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2021-10-20 (Actual); Primary Completion 2022-04-19 (Actual); Study Completion 2022-04-19 (Actual)

PRIMARY OUTCOMES:
Safety as assessed by adverse events (AEs) | From dosing (DTRI-031 or placebo) to final visit (Day 28)
  Incidence of treatment-emergent AEs

SECONDARY OUTCOMES:
Pharmacokinetics as measured by DTRI-031 plasma levels | From dosing to 24 hours after dosing
  Plasma concentration of DTRI-031 (after single dose of drug)
Plasma von Willebrand Factor (vWF) levels | From dosing to 24 hours after dosing
  Level of vWF following single administration of drug
Platelet Function | From dosing to 24 hours after dosing
  Whole blood platelet function closure times

CONTACTS AND LOCATIONS:
Locations (1):
- Nucleus Network, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No